CLINICAL TRIAL: NCT03973593
Title: Evaluation of Dynamics of Contraceptive Use, Discontinuation and Method Switching in Migori and Kitui Counties, Kenya
Status: Completed | Type: Observational
Sponsor: Jhpiego (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 00009062
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Family Planning; Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Enhancing contraceptive counseling on method continuation and switching — Health care workers and Community Health Volunteers will be trained on a contraceptive counseling package that enhances information on method continuation and switching. This will be done in the ten intervention facilities prior to enrollment of clients into the cohort study.

SUMMARY:
Kenya has made tremendous strides in improving contraceptive prevalence rate for the last 20 years, however the rate of contraceptive discontinuation as remained almost constant at 1 out of 3 women using a family planning method. Contraceptive discontinuation increases unmet need of family planning. Hence understanding the underlying reasons for discontinuation helps in designing programs that improve method satisfaction.

The primary goal of the study is to understand the factors leading to contraceptive discontinuation and switching among women of reproductive age (15 - 49 years) in Migori and Kitui counties, Kenya. The secondary goal is to assess whether a client-centered intervention focusing on contraceptive counseling can reduce modern contraceptive discontinuation and increase client satisfaction with use of modern contraceptive methods among women of reproductive age in the two counties.

The specific objectives are to:

1. To assess the quality of family planning services offered in health facilities in Migori and Kitui counties, Kenya
2. To explore describe barriers and facilitators of modern contraceptive discontinuation and method switch among women of reproductive age in Migori and Kitui counties.
3. To assess the client-centered intervention focusing on contraceptive counseling in reducing contraceptive discontinuation among women of reproductive age in Migori and Kitui counties, Kenya

DETAILED DESCRIPTION:
The 24 month prospective cohort study will seek to understand reasons for contraceptive discontinuation among women of reproductive age including adolescents in Kitui and Migori Counties, Kenya. The study will be implemented to assess determinants of contraceptive discontinuation after the barrier of lack of adequate counseling is removed. The barrier will be addressed by implementing an intervention focusing on a client-centered counseling approach in reducing contraceptive discontinuation among women accepting a contraceptive method. Ten health facilities with a high family planning caseload will be enrolled into the study. Counseling sessions will be conducted at the facilities using three channels:

1. Counseling by Community Health Volunteers (CHVs) The proposed intervention will identify CHVs and build their capacity on contraception with an aim of having them providing FP counseling and services in high volume facilities - thus providing additional human resources. Their current training on family planning focuses on general information for each contraceptive method but lacks adequate content on counseling for family planning. The CHV training package will be enhanced with additional content on contraceptive methods that will equip them with the necessary skills on counseling. They will also be trained on adolescent focused counseling as well. Once trained, the CHVs will offer counseling for family planning at facility level. Following the counseling, CHVs will provide a method including pills and injectables to women and girls who have come for a revisit, unless they request for contact with the health care worker. This is in line with the Kenya's Ministry of Health task sharing policy and family planning guidelines that allows CHVs to conduct community distribution of pills, condoms and injectables.
2. Individualized Counseling by Health Care Workers Once counseling has been done by the CHVs, the heath care workers will attend to the women in need for additional counseling and a method that the CHVs were unable to provide, for instance LARCs. The current counseling method used by the health care worker is the Balanced Counseling Strategy, which is cumbersome as it has a lot of information that overwhelms the providers and clients. The study proposes to adopt the counseling for continuation materials that will used to develop a simplified job aid for use by heath care workers to provide individualized counseling.
3. Partner Counseling by Health Care Workers (HCWs) CHVs will mobilize potential couples to jointly attend contraceptive counseling sessions by the health care workers. The health care workers will be trained on how to conduct couple counseling. Existing couples counseling materials will be adapted based on the information gathered from the formative assessment. The facility will identify a package of additional non-contraceptive related services for the men who will have accompanied their spouses for family planning services.

The investigators will enroll 1016 women of reproductive age in the following sub groups; Implant, IUD, Injectables and Pill users. Follow up interviews at 3, 6, and 12 months will be done to establish contraceptive use, discontinuation and method switching among women.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age (15-49 years) taking up a contraceptive method in the participating study facilities during the study enrollment period
2. A resident of the selected study region
3. Has access to a phone that they control for follow-up
4. Willing to be followed up to a period of 24 months after enrollment; four contacts.

Exclusion Criteria:

1. Women of reproductive age taking up a condom as their primary FP method, sterilization or an emergency contraceptive method
2. Participants not willing to consent
3. No access to phone

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women of reproductive age 15-49 years receiving a contraceptive method in the intervention facilities as new users to either the method or family planning
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Contraceptive discontinuation rate among FP users | up to 12 months
  The rate of contraceptive discontinuation among the prospective cohort FP users. Discontinuation will be of the baseline contraceptive method that the woman has initiated.

SECONDARY OUTCOMES:
Proportion of women reporting satisfaction with the quality of FP services offered at baseline | 12 months
  Proportion of women reporting extremely satisfied and satisfied with the information and services received at the health facility during initiation of contraception. Information will be collected from the baseline questionnaire to assess relationship between women reporting discontinuation and level of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Gathari Ndirangu, ObGyn, Study Director — Jhpiego
Locations (2):
- Kenya (2):
  - Kitui County Health facilities, Kitui
  - Migori County facilities, Migori

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol will be shared through publication in a peer-reviewed journal.
  De-identified participant data will be submitted to a data repository in accordance with the USAID policy where other researchers will have access.

REFERENCES:
- [Derived] Ontiri S, Mutea L, Muganda M, Mutanda P, Ajema C, Okoth S, Orero S, Odhiambo R, Biesma R, Stekelenburg J, Kabue M. Protocol for a prospective mixed-methods longitudinal study to evaluate the dynamics of contraceptive use, discontinuation, and switching in Kenya. Reprod Health. 2019 Sep 5;16(1):134. doi: 10.1186/s12978-019-0797-3. PMID 31488170